CLINICAL TRIAL: NCT02345005
Title: Multi-centre, Observational, Post-market, Real World Registry to Assess Outcomes of Patients Treated With the Gore® EXCLUDER® ILIAC BRANCH Endoprosthesis
Brief Title: Iliac Branch Excluder ReGistry (IceBERG)
Acronym: IceBERG
Status: Completed | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Collaborators: W.L.Gore & Associates (Industry)
Responsible Party: Principal Investigator, Michel Reijnen, Vascular surgeon, Rijnstate Hospital
Other Study IDs: 1060-011014
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Abdominal Aortic Aneurysms; Common Iliac Aneurysms; Aneurysm
Keywords: Vascular diseases; Aneurysm; Treatment Efficacy; Medical device; Population Register
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: The Gore® EXCLUDER® ILIAC BRANCH Endoprosthesis. — The Gore IBE device is a newly designed iliac branched device, that is used in combination with the widely accepted C3 Excluder endograft, for the exclusion of common iliac aneurysms and aorto-iliac aneurysms.

SUMMARY:
This post market registry consists of a retrospective and a prospective part. The first part is a retrospective registry of all implanted IBE devices of Gore in the Netherlands after CE mark was obtained, to get an initial insight on the feasibility and safety of this procedure. The second part is to prospectively register all data on implanted IBE Gore devices, in order to gain more robust data on the efficacy of the device in maintaining hypogastric artery patency.

DETAILED DESCRIPTION:
Rationale: The Gore IBE device is a newly designed iliac branched device, that is used in combination with the widely accepted C3 Excluder endograft for the exclusion of common iliac aneurysms and aorto-iliac aneurysms. The later has a proven safety and efficacy in excluding abdominal aortic aneurysms. The Gore IBE device got CE mark on October 2013. Technical and clinical data at short and long terms are still to be collected to give insight into technical success rates, patency data and long term follow-up.

Objective and design: This investigator-initiated post market registry consists of a retrospective and a prospective part. The first part is a retrospective registry of all implanted IBE devices of Gore in the Netherlands after CE mark was obtained, to get an initial insight on the feasibility and safety of this procedure. The second part is to prospectively register all data on implanted IBE Gore devices, in order to gain more robust data on the efficacy of the device in maintaining hypogastric artery patency.

Study population: All patients in whom a Gore IBE was or will be implanted. In the retrospective part of the study all implantations in the Netherlands will be gathered, whereas the prospective part will be expanded in Europe.

Main study parameters/endpoints: Aneurysm exclusion and reinterventions will be end-points of this study. As safety and feasibility is the main outcome of the retrospective part, the data will be analyzed at 30-days. Patients in the prospective study will be followed for 5 years, with the primary end-point being hypogastric side branch patency at 1-year. Clinical endpoints include freedom from symptoms of pelvic ischemia (buttock claudication, impotence and bowel ischemia) and freedom from aneurysm rupture.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Since this is a registry study, no burden or risk exist for the patient. There is also no direct benefit for the participating patients, but the gathered data will improve insight for patients with the same disease and might improve health care in the future for this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Provided written informed consent for data release
* Elective procedure; Indication for aorto-iliac endovascular stent graft repair, as determined by the treating physician

Exclusion Criteria:

* Patient is participating in another clinical study (RCT; interfering with endpoints)
* Patient's life expectancy <2 years as judged by the investigator
* Patient has a psychiatric or other condition that may interfere with the study
* Patient has a known allergy to any device component (ePTFE, FEP, nitinol)
* Patients with a systemic infection who may be at increased risk of endovascular graft infection
* Patient has a coagulopathy or uncontrolled bleeding disorder
* Patient has a ruptured, leaking, or mycotic aneurysm
* Patient had a CVA or an MI within the prior three months
* Patient is pregnant (Female patients of childbearing potential only)
* Other stents placed in CIA or hypogastric arteries than the Gore® EXCLUDER® iliac branch Endoprosthesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients in whom a Gore IBE was or will be implanted.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2025-07 (Actual); Study Completion 2025-07 (Actual)

PRIMARY OUTCOMES:
Safety and feasibility of the IBE device | Procedure and up to 30 days post procedure
  Primary endpoint of the retrospective part of the registry:
  - Safety and feasibility of the Gore IBE implantation up to 30 days, defined as immediate technical success; and complications from procedure up to 30 days
Primary patency of the hypogastric side branch | Up to 1 year postprocedure
  Primary endpoint of the prospective part of the registry: Primary patency of the hypogastric side branch at 1 year, and successful exclusion of the aneurysm without type I or II endoleak.

SECONDARY OUTCOMES:
Primary-assisted patency of the hypogastric branch | Measured at 1 month, 6 months, 1 year and then yearly up to 5 years
  Primary-assisted patency of the hypogastric branch measured with duplex ultrasound or CT during follow-up
Secondary patency of the hypogastric branch | Measured at 1 month, 6 months, 1 year and then yearly up to 5 years
  Secondary patency of the hypogastric branch measured with duplex ultrasound or CT
Buttock claudication | Measured at 1 month, 6 months, 1 year and then yearly up to 5 years
  Buttock claudication measured during regular follow-up
Erectile dysfunction | Measured at 1 month, 6 months, 1 year and then yearly up to 5 years
  Erectile dysfunction measured during regular follow-up and with the IIEF-5 questionnaire
Bowel ischemia | Measured at 1 month, 6 months, 1 year and then yearly up to 5 years
  Bowel ischemia measured following adverse events
Failure of the IBE device | Measured at 1 month, 6 months, 1 year and then yearly up to 5 years
  Freedom from type I and type III endoleak
Freedom from aneurysm rupture | Measured at 1 month, 6 months, 1 year and then yearly up to 5 years
  Aneurysm rupture will be measured following adverse events and reinterventions
Mortality | Measured at 1 month, 6 months, 1 year and then yearly up to 5 years
  Mortality measured during regular follow-up and adverse events
Patency | Measured yearly up to 5 years
  Patency of the hypogastric branch measured with duplex ultrasound or CT

CONTACTS AND LOCATIONS:
Overall Officials: Michel Reijnen, Principal Investigator — Rijnstate Hospital; Steven van Sterkenburg, Study Director — Rijnstate Hospital
Locations (8):
- Italy (3):
  - Fondazione Poliambulanza, Brescia
  - Cardarelli Hospital, Naples
  - San Filippo Neri Hospital, Rome
- Netherlands (2):
  - Rijnstate Hospital, Arnhem, Gelderland
  - Elisabeth Hospital, Tilburg
- Auckland Hospital, Auckland, New Zealand
- Spain (2):
  - Complexo Hospitelario Universitario de Ourense (CHUO), Ourense
  - Hospital Casa de Salud, Valencia

REFERENCES:
- [Background] Blankensteijn JD, de Jong SE, Prinssen M, van der Ham AC, Buth J, van Sterkenburg SM, Verhagen HJ, Buskens E, Grobbee DE; Dutch Randomized Endovascular Aneurysm Management (DREAM) Trial Group. Two-year outcomes after conventional or endovascular repair of abdominal aortic aneurysms. N Engl J Med. 2005 Jun 9;352(23):2398-405. doi: 10.1056/NEJMoa051255. PMID 15944424
- [Background] EVAR trial participants. Endovascular aneurysm repair versus open repair in patients with abdominal aortic aneurysm (EVAR trial 1): randomised controlled trial. Lancet. 2005 Jun 25-Jul 1;365(9478):2179-86. doi: 10.1016/S0140-6736(05)66627-5. PMID 15978925
- [Background] Prinssen M, Verhoeven EL, Buth J, Cuypers PW, van Sambeek MR, Balm R, Buskens E, Grobbee DE, Blankensteijn JD; Dutch Randomized Endovascular Aneurysm Management (DREAM)Trial Group. A randomized trial comparing conventional and endovascular repair of abdominal aortic aneurysms. N Engl J Med. 2004 Oct 14;351(16):1607-18. doi: 10.1056/NEJMoa042002. PMID 15483279
- [Background] Greenhalgh RM, Brown LC, Kwong GP, Powell JT, Thompson SG; EVAR trial participants. Comparison of endovascular aneurysm repair with open repair in patients with abdominal aortic aneurysm (EVAR trial 1), 30-day operative mortality results: randomised controlled trial. Lancet. 2004 Sep 4-10;364(9437):843-8. doi: 10.1016/S0140-6736(04)16979-1. PMID 15351191
- [Background] Brunkwall J, Hauksson H, Bengtsson H, Bergqvist D, Takolander R, Bergentz SE. Solitary aneurysms of the iliac arterial system: an estimate of their frequency of occurrence. J Vasc Surg. 1989 Oct;10(4):381-4. doi: 10.1067/mva.1989.13733. PMID 2795762
- [Background] Richardson JW, Greenfield LJ. Natural history and management of iliac aneurysms. J Vasc Surg. 1988 Aug;8(2):165-71. PMID 3294450
- [Background] Armon MP, Wenham PW, Whitaker SC, Gregson RH, Hopkinson BR. Common iliac artery aneurysms in patients with abdominal aortic aneurysms. Eur J Vasc Endovasc Surg. 1998 Mar;15(3):255-7. doi: 10.1016/s1078-5884(98)80186-x. PMID 9587341
- [Background] Hobo R, Sybrandy JE, Harris PL, Buth J; EUROSTAR Collaborators. Endovascular repair of abdominal aortic aneurysms with concomitant common iliac artery aneurysm: outcome analysis of the EUROSTAR Experience. J Endovasc Ther. 2008 Feb;15(1):12-22. doi: 10.1583/07-2217.1. PMID 18254666
- [Background] Timaran CH, Lipsitz EC, Veith FJ, Chuter T, Greenberg RK, Ohki T, Nolte LA, Snyder SA; Zenith Investigators. Endovascular aortic aneurysm repair with the Zenith endograft in patients with ectatic iliac arteries. Ann Vasc Surg. 2005 Mar;19(2):161-6. doi: 10.1007/s10016-004-0157-8. PMID 15776309
- [Background] Ziegler P, Avgerinos ED, Umscheid T, Perdikides T, Erz K, Stelter WJ. Branched iliac bifurcation: 6 years experience with endovascular preservation of internal iliac artery flow. J Vasc Surg. 2007 Aug;46(2):204-10. doi: 10.1016/j.jvs.2007.04.015. Epub 2007 Jun 27. PMID 17600664
- [Background] Abraham CZ, Reilly LM, Schneider DB, Dwyer S, Sawhney R, Messina LM, Chuter TA. A modular multi-branched system for endovascular repair of bilateral common iliac artery aneurysms. J Endovasc Ther. 2003 Apr;10(2):203-7. doi: 10.1177/152660280301000207. PMID 12877600
- [Background] Su WT, Stone DH, Lamparello PJ, Rockman CB. Gluteal compartment syndrome following elective unilateral internal iliac artery embolization before endovascular abdominal aortic aneurysm repair. J Vasc Surg. 2004 Mar;39(3):672-5. doi: 10.1016/j.jvs.2003.09.020. PMID 14981467
- [Background] Razavi MK, DeGroot M, Olcott C 3rd, Sze D, Kee S, Semba CP, Dake MD. Internal iliac artery embolization in the stent-graft treatment of aortoiliac aneurysms: analysis of outcomes and complications. J Vasc Interv Radiol. 2000 May;11(5):561-6. doi: 10.1016/s1051-0443(07)61606-6. PMID 10834485
- [Background] Karch LA, Hodgson KJ, Mattos MA, Bohannon WT, Ramsey DE, McLafferty RB. Adverse consequences of internal iliac artery occlusion during endovascular repair of abdominal aortic aneurysms. J Vasc Surg. 2000 Oct;32(4):676-83. doi: 10.1067/mva.2000.109750. PMID 11013030
- [Background] Yano OJ, Morrissey N, Eisen L, Faries PL, Soundararajan K, Wan S, Teodorescu V, Kerstein M, Hollier LH, Marin ML. Intentional internal iliac artery occlusion to facilitate endovascular repair of aortoiliac aneurysms. J Vasc Surg. 2001 Aug;34(2):204-11. doi: 10.1067/mva.2001.115380. PMID 11496269
- [Background] Mehta M, Veith FJ, Ohki T, Cynamon J, Goldstein K, Suggs WD, Wain RA, Chang DW, Friedman SG, Scher LA, Lipsitz EC. Unilateral and bilateral hypogastric artery interruption during aortoiliac aneurysm repair in 154 patients: a relatively innocuous procedure. J Vasc Surg. 2001 Feb;33(2 Suppl):S27-32. doi: 10.1067/mva.2001.111678. PMID 11174809
- [Background] Bratby MJ, Munneke GM, Belli AM, Loosemore TM, Loftus I, Thompson MM, Morgan RA. How safe is bilateral internal iliac artery embolization prior to EVAR? Cardiovasc Intervent Radiol. 2008 Mar-Apr;31(2):246-53. doi: 10.1007/s00270-007-9203-6. Epub 2007 Oct 24. PMID 17957407
- [Background] Rayt HS, Bown MJ, Lambert KV, Fishwick NG, McCarthy MJ, London NJ, Sayers RD. Buttock claudication and erectile dysfunction after internal iliac artery embolization in patients prior to endovascular aortic aneurysm repair. Cardiovasc Intervent Radiol. 2008 Jul-Aug;31(4):728-34. doi: 10.1007/s00270-008-9319-3. Epub 2008 Mar 13. PMID 18338212
- [Background] Torsello G, Schonefeld E, Osada N, Austermann M, Pennekamp C, Donas KP. Endovascular treatment of common iliac artery aneurysms using the bell-bottom technique: long-term results. J Endovasc Ther. 2010 Aug;17(4):504-9. doi: 10.1583/10-3112.1. PMID 20681766
- [Background] Karthikesalingam A, Hinchliffe RJ, Holt PJ, Boyle JR, Loftus IM, Thompson MM. Endovascular aneurysm repair with preservation of the internal iliac artery using the iliac branch graft device. Eur J Vasc Endovasc Surg. 2010 Mar;39(3):285-94. doi: 10.1016/j.ejvs.2009.11.018. Epub 2009 Dec 3. PMID 19962329
- [Background] Parlani G, Verzini F, De Rango P, Brambilla D, Coscarella C, Ferrer C, Cao P. Long-term results of iliac aneurysm repair with iliac branched endograft: a 5-year experience on 100 consecutive cases. Eur J Vasc Endovasc Surg. 2012 Mar;43(3):287-92. doi: 10.1016/j.ejvs.2011.12.011. Epub 2012 Jan 10. PMID 22240335
- [Background] Verzini F, Parlani G, Romano L, De Rango P, Panuccio G, Cao P. Endovascular treatment of iliac aneurysm: Concurrent comparison of side branch endograft versus hypogastric exclusion. J Vasc Surg. 2009 May;49(5):1154-61. doi: 10.1016/j.jvs.2008.11.100. PMID 19394544
- [Background] Verhoeven EL, Oikonomou K, Mohner B, Renner H, Ritter W; European C3 Global Registry Participants. First experience with the new repositionable C3 excluder stent-graft. J Cardiovasc Surg (Torino). 2011 Oct;52(5):637-42. Epub 2011 Jul 29. PMID 21799475
- [Background] Bastos Goncalves F, Jairam A, Voute MT, Moelker AD, Rouwet EV, ten Raa S, Hendriks JM, Verhagen HJ. Clinical outcome and morphologic analysis after endovascular aneurysm repair using the Excluder endograft. J Vasc Surg. 2012 Oct;56(4):920-8. doi: 10.1016/j.jvs.2012.03.263. Epub 2012 Jun 15. PMID 22703975
- [Background] Pratesi C, Piffaretti G, Pratesi G, Castelli P; ITalian Excluder Registry Investigators. ITalian Excluder Registry and results of Gore Excluder endograft for the treatment of elective infrarenal abdominal aortic aneurysms. J Vasc Surg. 2014 Jan;59(1):52-7.e1. doi: 10.1016/j.jvs.2013.06.067. Epub 2013 Sep 20. PMID 24055513